CLINICAL TRIAL: NCT06190262
Title: Community Based Group Psychoeducation for Relatives of Individuals With Mental Illness: A Feasibility Study
Brief Title: Community Based Group Psychoeducation for Relatives of Individuals With Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); OPEN, Open Patient data Explorative Network, Odense University Hospital, Region of Southern Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OP_1919; S-20232000 - 66 (Other: Videnskabsetisk Komitte); 23/25502 (Other: Internal Registry); 23/70733 (Other: Research Ethics Committee, University of Southern Denmark)
Record Dates: First submitted 2023-07-28; First posted 2024-01-05 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Caregiver Burden; Caregiver Burnout; Well-Being, Psychological; Coping Strategies; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Caregiver Burden; Psychological Well-Being; Behavior

STUDY DESIGN:
Intervention Model Description: One arm pre-test/post-test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychoeducation (Experimental): The experimental condition consists of a psychoeducation program with six sessions. Two of the sessions are online. A teacher and a volunteer will lead the sessions. The topic of the sessions are diverse and cover topics such as mental illness, the diathesis-stress model, treatment of mental illness, caregiver coping mechanisms and caregiver rights.
  Before the first session, participants are asked to fill in an online questionnaire with background information and well-being indicators. After the last session, participants are asked to fill in another short questionnaire with the same well-being indicators and also a measure of their satisfaction with the program.
  Interventions: Behavioral: The intervention is community based group psychoeducation

INTERVENTIONS:
Behavioral: The intervention is community based group psychoeducation — The intervention is community based group psychoeducation

SUMMARY:
The goal of this one-arm pre-test/post-test study is to evaluate the feasibility and preliminary effect of a community-based psychoeducational group intervention for informal caregivers of individuals with mental illness.

The main questions it aims to answer are:

* What is the feasibility and acceptability of the intervention?
* What is the preliminary effect of the intervention?

Participants self-select to the intervention and participation in the evaluation is voluntary. Participants will be asked to:

* Answer a questionnaire before and after their participation
* Some participants will be invited for an in-depth interview

There is no comparison group, but feasibility and acceptability will also be explored by asking the implementation team (e.g. project leaders and teachers) to participate in:

* In-depth interviews
* Answering shorter questionnaires about provider acceptability

DETAILED DESCRIPTION:
The program/intervention:

The group-based psychoeducational program focuses on enhancing informal caregivers' or relatives' understanding of their loved ones' mental illnesses and equips them with coping strategies. The main goal is to improve caregivers' knowledge of mental illnesses and their ability to navigate in their daily life/their role as an informal caregiver without becoming overburdened.

The specific program was collaboratively developed by a non-government organization and the regional psychiatry in one of Denmarks five Regions. Participants self-select to the program and participation is free of cost.

The program consists of six sessions, two of which are conducted online. The program is designed for groups of 16-20 individuals.

Session 1: The first session serves as an introduction to the program, where participants get acquainted with each other and familiarize themselves with the program's content. During this session, participants are encouraged to establish their own rules while also discussing the "Chatham House rules."

Session 2: Moving on to the second session, the focus is on disseminating knowledge about mental illnesses, treatment, and the distinctions between regional psychiatry and community-based treatments. A compassion-focused exercise is also included during this session.

Session 3: The third session centers on providing information about various treatment opportunities, exploring different types of treatment in addition to medication and talk therapy. Moreover, participants gain insights into how they can be involved in the treatment process if the patient provides their consent. This session is conducted online.

Session 4: The fourth session delves into the caregiver role and self-care strategies. Participants are introduced to different coping-strategies.

Session 5: In the fifth session, the focus shifts to the rights of the participants, such as their entitlement to care days and information about other caregiver interventions in the community. This session is conducted online.

Session 6: Finally, in the last session, all the topics covered throughout the program are summarized, and support groups are established to provide ongoing assistance and encouragement.

In 2024, around 24 courses will be offered, each spanning a duration of 35-70 days. The sessions will be conducted. The sessions will be scheduled either weekly (with 6 sessions over a 35-day period) or bi-weekly (with 6 sessions over a 70-day period).

The evaluation:

All participants in the program will be asked to participate in the evaluation. Participation in the evaluation is completely voluntary.

The primary purpose of the evaluation is to use the results of the evaluation to continuously revise the program to reflect the needs of the participants. By the end of 2025, the program will have undergone the last revision, and be ready to move on to a full evaluation using a RCT design. Thus, in line with guidance from the UK Medical Council Research Framework (MRC) and the National Institute of Health Research framework, the present study is an initial step in determining if the developed intervention is feasible and acceptable for relatives to individuals with mental illness. A mixed-methods approach was chosen to explore indications of participants' response and view to the intervention and thereby gain a more full understanding of the intervention acceptability and feasibility.

The principal aims of this study are as follows:

1. To assess the feasibility and acceptability of the intervention, the investigators aim to:

   1. Quantify recruitment rate and attendance rate
   2. Measure participants' satisfaction with the intervention
   3. Qualitatively explore participants satisfaction and their ideas for development
   4. By using purposeful sampling strategies, some participants will be invited to take part in an in-depth interview about their experience with the program and about their perspective on facilitators and barriers of the intervention. They will also be asked about how to improve the program in the future.
2. To assess the preliminary effectiveness of the intervention, participants are asked to:

   1. Self-report on their well-being before and after the intervention
   2. Self-report on their level of burnout before and after the intervention
   3. Self-report on their level of resilient coping before and after the intervention

   This evidence will provide an initial indication of whether the intervention can contribute to change within this group. Estimated effect sizes will provide the parameters for a definitive randomized controlled trial. Data will be explored using the reliable and clinically significant change analysis. This analysis allows pre- and post-treatment scores to be compared to see if participants have achieved a level of difference that could be categorized as real and not due to measurement error. Furthermore this score can be helpful to determine if the change seen is clinically significant.
3. To assess feasibility and acceptability from the providers, the investigators aim to:

   1. Conduct in-depth interviews with members of the implementation teams (such as project leaders and teachers in the program).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to read, speak, and understand the Danish langugage
* Relative/informal caregiver of an individual with a mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Recruitment rate is monitored throughout the study period (1 year)
  To measure the feasibility of the intervention, there is a measure of recruitment rate (number of participants recruited/time period in months).
Attendance rate | Attendance rates are monitored throughout the study period (1 year)
  To measure feasibility of the intervention, there is a measure of attendance rate: (number of participants attending/total number of enrolled participants) * 100
Retention rate | Retention rates are monitored throughout the study period (1 year)
  To measure feasibility of the intervention, there is a measure of retention rate: (number of participants remaining/intital Number of Enrolled Participants) * 100
Satisfaction, quantitative measure | Immediatly after participants finish the last session (session six, either 35 days or 70 days after enrolling in the intervention).
  To measure acceptability of the intervention, participants' overall satisfaction with the program will be measured. This measure is based on 11 questions, that are rated on a 4-point Likert-Scale. Higher scores indicate higher satisfaction.
Satisfaction, qualitative measure | Immediatly after participants finish the last session (session six, either 35 days or 70 days after enrolling in the intervention).
  To measure acceptability of the intervention, participants are invited to write about their experience with the program and their ideas for program development.
Suitability, qualitative measure | Individual semi-structured interviews will be conducted throughout the study period (1 year).
  Based on individual semi-structured interviews with some of the participants the investigators will evaluate whether the intervention fits the target population's needs, preferences, and cultural context. This measure will be used to assess whether any modifactions are needed to enhance the programme suitability.
Barriers and facilitators, qualitative measure (provider perspective) | Focus-group interviews will be conducted throughout the study period (1 year).
  Based on focus-group interviews with the teachers and other stakeholders, qualitative data will be collected to understand the providers' experiences, perceptions, and suggestions for improvement of the program.

SECONDARY OUTCOMES:
Well-being: WHO-5 well-being index | 1 week before the first session, and immediatly after the last session (session six, either 35 days or 70 days after enrolling in the intervention).
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing. It is composed of five questions that are rated on a 6-point Likert-Scale, where 5 = all the time and 0 = at no time. The raw score ranging from 0 to 25 is multiplied by 4 to give the final score from 0 (representing the worst imaginable well-being) to 100 (representing the best imaginable well-being).
Personal Burnout: Copenhagen Burnout Inventory (CBI; personal burnout) | 1 week before the first session, and immediatly after the last session (session six, either 35 days or 70 days after enrolling in the intervention).
  The CBI consists of three inventories measuring 1) personal burnout, 2) work-related burnout, and 3) client-related burnout, for use in different domains. In this study, only the personal burnout inventory is used. The personal burnout inventory consists of six questions that are rated on a 5-point Likert-Scale ranging from 1 (never/almost never), 2 (seldom), 3 (sometimes), 4 (often), and 5 (always).
  Total score on the scale is the average of the scores on the items, and higher scores indicate higher levels of burnout.
Coping: Brief resilient coping scale | 1 week before the first session, and immediatly after the last session (session six, either 35 days or 70 days after enrolling in the intervention).
  The Brief Resilient Coping Scale captures tendencies to cope with stress adaptively. The scale focuses on the tendency to effectively use coping strategies in flexible, committed ways to actively solve problems despite stressful circumstances. The four items are rated on a 5-point Likert-Scale ranging from 1 (does not describe me at all) to 5 (describes me very well). Higher scores indicate more resilient coping. The score ranges from 4 - 20. Scores from 4-13 represent low resilient copers; scores from 14-16 represent medium resilient copers; and scores from 17-20 represent high resilient copers.

OTHER OUTCOMES:
Relationship satisfaction | 1 week before the first session, and immediatly after the last session (session six, either 35 days or 70 days after enrolling in the intervention).
  Relationship satisfaction is measured using one item from the Couples Satisfaction Index. The question relates to the overall satisfaction with the relationship, and is measured on a 6-point Likert-Scale, ranging from 1 (not at all) to 6 (completely). Higher scores indicate higher satisfaction.
Self-reported teacher fidelity | through study completion, an average of 1 year
  To measure feasibility of the intervention, teacher adherence to the manual is measured. The teachers fill in a fidelity checklist, which consists of 4-6 items that measure the extent to which key components of the intervention were delivered. The questions are rated on a Likert-Scale ranging from 1 (not at all) to 3 (a lot).

CONTACTS AND LOCATIONS:
Overall Officials: Rikke Amalie Agergaard Jensen, Ph.d., Principal Investigator — Department of Regional Health Research, University of Southern Denmark
Locations (1):
- Center for Involvement of Relatioves, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study are not expected to be made available due to sensitive information.

REFERENCES:
- [Background] Sinclair VG, Wallston KA. The development and psychometric evaluation of the Brief Resilient Coping Scale. Assessment. 2004 Mar;11(1):94-101. doi: 10.1177/1073191103258144. PMID 14994958
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Funk JL, Rogge RD. Testing the ruler with item response theory: increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. J Fam Psychol. 2007 Dec;21(4):572-83. doi: 10.1037/0893-3200.21.4.572. PMID 18179329
- [Background] Morley S, Williams A, Hussain S. Estimating the clinical effectiveness of cognitive behavioural therapy in the clinic: evaluation of a CBT informed pain management programme. Pain. 2008 Jul 31;137(3):670-680. doi: 10.1016/j.pain.2008.02.025. Epub 2008 Apr 3. PMID 18394806